CLINICAL TRIAL: NCT04247451
Title: Diabetic Foot Surgery Patients: What is Their Metabolic Profile and Are Nutritional Goals Met
Acronym: DIM-SUUM
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: low inclusion rate
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Elisabeth De Waele, Head of Clinics ICU, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BUN 143201941164
Record Dates: First submitted 2020-01-08; First posted 2020-01-30 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Diabetic Foot Ulcer; Nutrition Disorders
MeSH Terms: conditions — Diabetic Foot; Nutrition Disorders | interventions — Metabolome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional group (Experimental): Nutritional intake: these data will be evaluated daily during preoperative hospitalization, at home, and during the actual hospitalization, from surgical intervention to discharge. Before the follow-up consultation, patients will keep a food diary. The dieticians will calculate intake and need.
  Metabolic data: body composition using BIA (Nutrilab Akern) and REE using indirect calorimetry (Cosmed Q NRG) will be analyzed in three timepoints: preoperative, postoperative and at follow-up consultation. This measurements take maximum ten minutes and do not cause discomfort to the participants.
  Interventions: Diagnostic Test: Metabolic profile and nutritional goals in diabetic foot surgery patients

INTERVENTIONS:
Diagnostic Test: Metabolic profile and nutritional goals in diabetic foot surgery patients — Nutritional intake: these data will be evaluated daily during preoperative hospitalization, at home, and during the actual hospitalization, from surgical intervention to discharge. Before the follow-up consultation, patients will keep a food diary. The dieticians will calculate intake and need.
  Metabolic data: body composition using Bio electrical Impedance Analysis BIA (Nutrilab Akern) and Resting Energy Expenditure REE using indirect calorimetry (Cosmed Q NRG) will be analysed in three timepoints: preoperative, postoperative and at follow-up consultation. This measurements take maximum ten minutes and do not cause discomfort to the participants.

SUMMARY:
Prospective interventional follow-up of diabetic foot surgery patients, their metabolic/nutritional profile, and the nutritional adequacy in the perioperative setting.

Primary objective: to establish the preoperative metabolic profile of diabetic patients scheduled for foot surgery and determine the postoperative nutritional status. The daily values of caloric intake compared to caloric need and protein intake compared to protein need will be evaluated as primary endpoint. [Actual daily caloric and protein intake is compared to the calculated need.] These values will each be presented as relative %.

Wound healing is an anabolic process that requires ample access to nutrients. Insulin is considered the main anabolic hormone of the body, and regulates the metabolism of carbohydrates, fats and proteins. Diabetic patients lack this very hormone, and in addition are required to follow a strict dietary regime that further limits caloric and protein intake. Very little research had been done to evaluate the role of malnutrition in delayed wound healing.

Overall: What is the metabolic/nutritional profile of a diabetes patient with foot wounds undergoing surgery? Is the intake of proteins and caloric adequate in the perioperative setting and are nutritional goals met? Is there a possibility for iatrogenic malnutrition? What kind of nutrition would possibly be useful to optimize intake?

DETAILED DESCRIPTION:
Diabetes mellitus is an important risk factor for foot ulcers often leading to minor or even major amputations, all with functional impairment.

The pathophysiology of diabetic foot wounds is multifactorial, and a combination of treatment modalities is required to accomplish wound healing. As such, infection control (by means of surgery as well as antibiotics), off-loading and revascularization all contribute to a successful outcome.

Wound healing invariably requires some degree of tissue regeneration, which is an anabolic process that requires ample access to nutrients and energy. In spite of malnutrition being detrimental to wound healing, the nutritional status of the diabetic foot patient is rarely taken into account when devising up a treatment regimen. This is remarkable, as diabetic patients are prone to inadequate energy intake because of three important reasons.

First, they lack insulin, which is considered the main anabolic hormone of the body. Insulin regulates the uptake, storage and conversion of several crucial nutrients, like carbohydrates, fats and proteins, and plays such a pivotal role in energy house holding that diabetes affects almost all cellular processes in the body. Second, diabetic patients are invariably put on a dietary regime in order to maintain strict glycemia control. This requires a patient to schedule meals at very regularly timed intervals, of consistent caloric quantity. In addition, dietary intake has to be adapted to prior or scheduled physical exercise. The primary objective of a diabetes diet being glycemia control may consequently mean that it falls short as an optimal regimen for wound healing.

Third, diabetic foot patients that undergo surgery frequently deviate from their customary diet. Fasting is often mandatory for anesthesia, and is usually prolonged due to neuropathic gastroparesis. Antibiotics may interfere with gastro-intestinal uptake. Hypermetabolic stress due to infection or surgery may temporarily increase energy expenditures.

Low-extremity ulcers are an important health issue, with an extended impact on patients and health. Nutrition as a therapeutic intervention is well established in several domains of medicine, such as the treatment of critically ill patients. A nutritional treatment can alter outcome, when performed in an individualised, patient-tailored setting.

In a randomized prospective way, the investigator's research group proved patient relevant outcome changes when an adequate nutritional therapy was applied: newly diagnosed cancer patients experienced significant less unplanned hospital admissions and saw a decline in the need of dose reduction of their anticancer treatment, as well as a rise in survival. A similar success was seen in a prospective intervention in patients planned for cardiac surgery: a program of close clinical monitoring and interventions by the use of dietary modifications, oral supplements or enteral or parenteral nutrition (or a combination thereof) resulted in a better survival of female patients and a lowered infection rate in male and female CABG and valve surgery patients. There were less episodes of postoperative arrhythmia, and the pneumonia rate went down.

ELIGIBILITY:
Inclusion criteria

* Age > 18years
* under oral or insulin therapy for diabetes mellitus
* patient recruitment at the multidisciplinary at the diabetic wound clinic of the University Hospital Brussel
* scheduled for surgery, with an indication related to the wound(s).

Exclusion criteria

* Presence of other metabolic diseases (inborn/acquired such as hyperthyroidism)
* Incapacity to undergo research investigations (relative CI to body composition measurement by Bio electrical impedance BIA: cardiac defibrillator)
* Limb- or life threatening disease
* Patient or relatives is/are unable to accurately record dietary intake

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficiency of nutritional therapy: Dietary intake (food diary; in Kcal) compared to caloric need (indirect calorimetry; Kcal) | an average of 3 weeks (perioperative period)
  Actual daily caloric and protein intake compared to the calculated need. These values will each be presented as relative %.

SECONDARY OUTCOMES:
Caloric needs (indirect calorimetry; Kcal) in diabetic foot surgery | an average of 3 weeks (perioperative period)
  resting energy expenditure measured by indirect calorimetry before and after surgery
Evaluation of choice for oral nutritional supplements, enteral nutrition and parenteral nutrition (%) | an average of 3 weeks (perioperative period)
  evaluation of nutritional possibilities by health care providers

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth De Waele, MD, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Brussels, Belgium